CLINICAL TRIAL: NCT02628223
Title: A Randomized Trial of 180 Degree vs. 360 Degree Selective Laser Trabeculoplasty as Initial Therapy for Glaucoma
Brief Title: 180 Degree vs. 360 Degree Selective Laser Trabeculoplasty as Initial Therapy for Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21921
Record Dates: First submitted 2015-11-23; First posted 2015-12-11 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension; Glaucoma, Open Angle, Pseudo-exfoliative; Pigment Dispersion Syndrome; Glaucoma
Keywords: glaucoma; Elevated IOP; Selective Laser Trabeculoplasty; SLT; open angle glaucoma; ocular hypertension; Glaucoma, Open Angle, Pseudo-exfoliative; pigment dispersion syndrome; Pseudoexfoliation; IOP ≥ 21 mmHg
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Glaucoma-Related Pigment Dispersion Syndrome | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 180 degrees (Active Comparator): 180 degrees of Selective Laser Trabeculoplasty using Neodymium:Yttrium Aluminum Garnet (YAG) laser
  Interventions: Procedure: Selective Laser Trabeculoplasty; Device: Neodymium:Yttrium Aluminum Garnet (YAG) laser
- 360 degrees (Active Comparator): 360 degrees of Selective Laser Trabeculoplasty using Neodymium:Yttrium Aluminum Garnet (YAG) laser
  Interventions: Procedure: Selective Laser Trabeculoplasty; Device: Neodymium:Yttrium Aluminum Garnet (YAG) laser

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — The procedure uses light energy provided by a neodymium (Nd):Yttrium Aluminum Garnet (YAG) laser that is directed into the iridocorneal angle via a goniolens viewed through a standard slit lamp.
  Other Names: SLT
Device: Neodymium:Yttrium Aluminum Garnet (YAG) laser — The procedure uses a 400 μm spot size of light energy provided by a low-energy, Q-switched, frequency-doubled (532 nm) neodymium (Nd):Yttrium Aluminum Garnet (YAG) laser with a short pulse duration of 3 nanoseconds that is directed into the iridocorneal angle via a goniolens viewed through a standard slit lamp.
  Other Names: Nd:YAG laser

SUMMARY:
Selective laser trabeculoplasty (SLT) is a well-recognized way to lower eye pressure in treatment of glaucoma. This treatment is performed for 180 degrees or 360 degrees, and studies at academic centers have shown mixed results when comparing the success rates of 180 degrees or 360 degrees. Both protocols are now typically done by comprehensive ophthalmologists. However, there is no data that compares success rates of 180 degrees and 360 degrees in the community setting.

DETAILED DESCRIPTION:
This study is designed as a prospective evaluation of the two treatment algorithms for SLT by measuring intraocular pressure (IOP) after treatment. The hypothesis is that 360 degrees of SLT will produce a greater reduction in IOP than 180 degrees of SLT at 3 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been diagnosed with open-angle glaucoma including ocular hypertension, pseudoexfoliation and pigment dispersion syndrome
* greater than 18 years of age
* initial intraocular pressure (IOP) of ≥ 21 mmHg

Exclusion Criteria:

* prior medical or laser therapy to lower IOP
* previous incisional glaucoma surgery before the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Henderer, MD, Principal Investigator — Temple University; Sophia Siu, MD, Study Director — Temple University
Locations (2):
- United States (2):
  - Brandywine Eye Center, Wilmington, Delaware
  - Levin Luminais Chronister Eye Associates, Thorndale, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 180 Degrees | 360 Degrees
Started | 38 | 38
Completed | 38 | 36
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 180 Degrees | 360 Degrees | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 29 | 33 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (8.6) | 71.9 (6.7) | 71.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 19 | 18 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 32 | 28 | 60
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1
Hypertension [Count of Participants; unit: Participants] | 25 | 29 | 54
Diabetes [Count of Participants; unit: Participants] | 9 | 14 | 23
Glaucoma (mild, moderate, severe, indeterminant) [Count of Participants; unit: Participants]
  Mild | 13 | 12 | 25
  Moderate | 4 | 8 | 12
  Severe | 1 | 2 | 3
  Indeterminant | 7 | 0 | 7
  No Glaucoma | 13 | 16 | 29
Ocular Hypertension [Count of Participants; unit: Participants] | 8 | 12 | 20
Pseudoexfoliation [Count of Participants; unit: Participants] | 6 | 1 | 7
Pigment Dispersion Syndrome [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) Measured by Tonometry in Millimeters of Mercury at Three Months of Follow-up
Description: Intraocular pressure (IOP) measured by tonometry in millimeters of mercury at three months of follow-up
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 180 Degrees | 360 Degrees
Number analyzed (Participants) | 38 | 36
mm Hg | 20.7 (5.4) | 19.1 (4.1)

2. Secondary Outcome: Intraocular Pressure (IOP) Measured by Tonometry in Millimeters of Mercury at 1 Year of Follow-up
Description: Intraocular pressure (IOP) measured by tonometry in millimeters of mercury at 1 year of follow-up
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 180 Degrees | 360 Degrees
Number analyzed (Participants) | 38 | 36
mm Hg | 18.7 (3.1) | 19.0 (4.4)

3. Secondary Outcome: Intraocular Pressure (IOP) Measured by Tonometry in Millimeters of Mercury at Time at Which Additional Glaucoma Therapy is Required
Description: Intraocular pressure (IOP) measured by tonometry in millimeters of mercury at time at which additional glaucoma therapy is required
Time Frame: within 1 year of study intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 180 Degrees | 360 Degrees
Number analyzed (Participants) | 38 | 36
mm Hg | 24.7 (4.0) | 23.7 (3.3)

4. Secondary Outcome: Intraocular Pressure (IOP) Measured by Tonometry in Millimeters of Mercury at Last Follow-up
Description: Intraocular pressure (IOP) measured by tonometry in millimeters of mercury at last follow-up
Time Frame: within 1 year of study intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 180 Degrees | 360 Degrees
Number analyzed (Participants) | 38 | 36
mm Hg | 18.2 (2.8) | 18.3 (4.9)

5. Other Pre Specified Outcome: Number of Participants With Intraocular Pressure (IOP) Spike Assessed by Tonometry
Description: If IOP spike occurs, it will be treated accordingly.
Time Frame: within 1 year of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | 180 Degrees | 360 Degrees
Number analyzed (Participants) | 38 | 36
Participants | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Trabeculitis Assessed by Ophthalmic Exam and Gonioscopy
Description: If trabeculitis occurs, it will be treated accordingly.
Time Frame: within 1 year of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | 180 Degrees | 360 Degrees
Number analyzed (Participants) | 38 | 36
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 180 Degrees | 360 Degrees
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/38 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 Degrees (N=38) | 360 Degrees (N=36)
Corneal Abrasian (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There were some limitations to this study that include: No standardized definition of who needed laser; No standardized technique other than the amount of meshwork lasered; No standardized IOP checking device; No standardized post op drop regimen; No standardized follow up interval.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT02628223/Prot_SAP_000.pdf